CLINICAL TRIAL: NCT05234060
Title: Study of People's Profile Living in France Who Could be Interested in the Use of a Nanohydroxyapatite Toothpaste
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0046
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Dental Caries; Hydroxyapatite
Keywords: Cariostatic Agents; Toothpaste
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nano-hydroxyapatite is an interesting candidate to be a substitute for fluor in toothpastes or a complement to fluorides in order to prevent caries. The objective of this transversal descriptive study is to evaluate the profiles of people living in France who could be interested in using a nano-hydroxyapatite based toothpaste.

Participants in this transversal descriptive study have been chosen by a self-administered method. Before answering 16 questions, the participants were asked to watch a short video describing the main concepts to know about fluoridated toothpastes and nano-hydoxyapatite toothpastes. Pros and cons of each one them were mentioned. In order to compare the answers, pivot tables have been produced.

ELIGIBILITY:
Inclusion criteria:

* Internet acces
* Interested in the Use of a Nanohydroxyapatite Toothpaste

Exclusion criteria:

* Age < 18 years
* Peoples who no lives in France

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peoples who lives in France
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Number of people interested in using toothpaste based on nano-hydroxyapatite | 1 day
  Number of people interested in using toothpaste based on nano-hydroxyapatite

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Giraudeau, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC